CLINICAL TRIAL: NCT05017454
Title: Assessment of Efficacy and Safety of Sodium Valproate -Loaded Nanospanlastics in Patients With Patchy Alopecia Areata in Comparison to Conventional Therapy With Topical Steroids: a Randomized Controlled Study, With Clinical, Dermoscopic and Molecular Asessements
Brief Title: Sodium Valproate-loaded Nanospanlastics in Patchy Alopecia Areata in Comparison to Topical Steroids
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, heba ahmed abdelgayed ibrahim, Dr, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 264199200
Record Dates: First submitted 2021-08-14; First posted 2021-08-23 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Alopecia Areata
Keywords: sodium valproate-loaded nanospanlastic; topical steroids; beta catenin; alopecia areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sodium valproate group (Experimental): Group 1 will be treated with the optimized sodium valproate-loaded nanospanlastic dispersion, twice daily on the affected areas of the scalp for 3 months
  Interventions: Drug: the optimized sodium valproate-loaded nanospanlastic dispersion
- topical steroid group (Active Comparator): Group 2 will be treated with the marketed mometasone furoate lotion twice daily on the affected areas of the scalp for 3 months
  Interventions: Drug: mometasone furoate lotion

INTERVENTIONS:
Drug: the optimized sodium valproate-loaded nanospanlastic dispersion — participants will apply the optimized sodium valproate-loaded nanospanlastic dispersion twice daily, on the affected areas of the scalp for 3 months
  Arms: sodium valproate group
Drug: mometasone furoate lotion — participants will apply marketed mometasone furoate lotion twice daily on the affected areas of the scalp for 3 months
  Arms: topical steroid group

SUMMARY:
the aim of this study is to assess the efficacy and safety of sodium valproate-loaded nanospanlastic in the treatment of patchy AA, in comparison to conventional therapy with topical steroids

DETAILED DESCRIPTION:
Alpopecia Areata (AA) is the second common cause of non-scarring hair loss, the disease has huge negative impact on patients' quality of life, social and psychological status. The underlying pathogenesis of AA is not fully characterized, Yet the collapse of immune privilege and generation of autoimmune attack against unknown follicular antigens are the most agreed-upon theories behind the disease. In spite of various therapeutic armamentariums available for AA, no single agent has been proven efficacious regarding reversing hair loss and establishing long-term response.

keeping in mind the burden of the disease together with lacking effective treatments, a need for further therapies is colossal.

Wnt-b catenin pathway is one of the crucial signalling pathways that regulate hair cycling. An increasing body of evidence is supporting the fact that wnt-b catenin pathway is inhibited in AA, and therefore contributing to the hair loss that characteize the disease.

Sodium valproate (SV), a well-known anti-epileptic drug, was found to inhibit Glycogen synthase kinase-3beta (GSK3β) in neuronal cells as one of the possible antiepileptic mechanisms of SV. GSK3B is a well-known inhibitor of β-catenin activity in dermal papilla cells (DPCs), and thus induces catagen-like changes in these cells. So the idea of using topical SV to promote hair regrowth via activation of b catenin came up and attracted the interests of investigators. recently an optimized sodium valproate-loaded nanospanlastics topical formula promisingly achieved clinical equivalence with 5% minoxidil lotion in AGA, with a superior safety profile to minoxidil

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate patchy alopecia areata, which is defined as less than 50% involvement of the entire scalp
* Age above 12 years.
* Both genders.
* Patients with patchy alopecia areata, with 2 patches or more

Exclusion Criteria:

* Patients having single patch alopecia areata (at least 2 patches are required, as one patch will be left untreated to exclude the possibility of spontaneous remission)
* Affection of more than 50% of the scalp area
* Patients with alopecia totalis or universalis
* Patients with ophiasis
* Age: Less than 12 years old.
* Pregnant or lactating females
* Patients with history of or existing scalp skin diseases, infections or skin cancer
* Severe systemic illness (as uncontrolled DM or hypertension, liver or renal diseases) and immune-compromised patients
* Patients with concomitant autoimmune diseases as suspected by history or confirmed by previous investigations
* Diagnosis or history of local dermatological disease in the scalp apart from AA such as eczema, seborrheic dermatitis, psoriasis.
* Any psychiatric illness or psychological state impairing future compliance or influencing expectations of the patient

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
- Treatment success | 6 months
  defined by achieving ≥ 50% reduction in baseline SALT score at end-of-study and/or achieving patient global assessment of improvement (PGAI) ≥ 50%.

SECONDARY OUTCOMES:
molecular Assessment of treatment success rate of SV-loaded nanospanlastics in the treatment of mild to moderate patchy AA in comparison to conventional therapy with topical steroids | 3 months
  Assessment of expression of both beta-catenin and Axin2 in lesional scalp of patients with patchy AA before and after treatment with sodium valproate-loaded nanospanlastics, in comparison to conventional therapy with topical steroids
Dermoscopic evaluation of hair regrowth | 3 months
  This evaluation will determine the number of dystrophic hairs in the patch area at baseline to be compared after the end of treatment. Markers for dystrophic hairs include exclamation-mark hairs, black dots, yellow dots and pigtail regrowing hair. The percentage of dystrophic hairs will be evaluated on a four-point scale: 3, > 50%; 2, 30-50%; 1, 1-29%; 0, no dystrophic hairs
Patient global assessment of improvement | 3 months
  Patient global assessment of improvement will be evaluated at the end of study, and will be scored as the following; (0 =no regrowth; 1 = <25% of regrowth; 2 = 25%-49% of regrowth; 3 = 50%-74% of regrowth; 4 = 75%-99% of re- growth; 5 = 100% of regrowth)
Clinical satisfaction of each patient | 3 months
  Clinical satisfaction of each patient will be made using a 10-point visual analogue scale (VAS, 0-10; the 0 level was defined as "Not satisfied at all," while a level of 10 was defined as "completely satisfied")
Subjective assessment of any encountered adverse effects | 3 months
  Subjective assessment of any encountered adverse effects (burning, itching) will also be performed. This will be determined on a four-point scale: 3, strong sensation; 2, moderate sensation; 1, mild sensation; 0, no itching or burning sensation
Patient satisfaction regarding characteristics of the used topical treatment | 3 months
  Patient satisfaction regarding characteristics of the used topical treatment, for example (texture, spreadability, hair matting, odour). This will be evaluated on a 3-point scale; 0=unsatisfied, 1=moderately satisfied, 2=extremely satisfied
Dermatology Life Quality Index (DLQI) | 3 months
  Dermatology Life Quality Index (DLQI) will be evaluated at baseline and at the end of therapy, using a validated DLQI questionaire
Assessment of relapse | 6 months
  Patients who achieved 100% reduction in baseline SALT after 3 months of treatment (end of therapy) were followed up for additional 3 months (end of study) to monitor any relapses.

CONTACTS AND LOCATIONS:
Overall Officials: heba ahmed, Msc in dermatolo, Principal Investigator — Kasralainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Kasralainy Hospital, Dermatology Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mogawer RM, Fawzy MM, Mourad A, Ahmed H, Nasr M, Nour ZA, Hafez V. Topical sodium valproate-loaded nanospanlastics versus conventional topical steroid therapy in alopecia areata: a randomized controlled study. Arch Dermatol Res. 2024 Jan 3;316(2):64. doi: 10.1007/s00403-023-02785-1. PMID 38170256